CLINICAL TRIAL: NCT00024141
Title: 5-Flourouracil Preceded by Irinotecan In Patients With Advanced Solid Tumors: A Pilot Study
Brief Title: Irinotecan Followed by Fluorouracil in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Patrick Creaven, MD, Institutional Review Board
Purpose: Treatment
Other Study IDs: CDR0000068895; RPCI-RP-01-01
Record Dates: First submitted 2001-09-13; First posted 2003-06-20 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of irinotecan followed by fluorouracil in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the optimal dose of irinotecan when administered before fluorouracil in patients with advanced solid tumors.
* Determine the toxic effects of this regimen in these patients.
* Correlate the pharmacokinetics of irinotecan with its biologic effects in these patients.
* Assess, in a preliminary manner, the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose de-escalation study of irinotecan.

Patients receive irinotecan IV over 90 minutes on days 1, 8, 15, and 22 and fluorouracil IV over 5 minutes on days 2, 9, 16, and 23. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive decreasing doses of irinotecan until the optimal dose is determined. The optimal dose is defined as the dose at which at least 3 of 6 patients show evidence of recruitment of cells into the S phase at 24 hours after irinotecan administration.

PROJECTED ACCRUAL: A total of 18-24 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent or metastatic solid tumor that is not amenable to curative surgery, radiotherapy, or conventional chemotherapy of proven value
* Must have disease that can be safely and readily biopsied under local anesthesia (including, but not limited to, subcutaneous metastases, superficial lymph node metastases, or ascites)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST less than 2 times ULN
* Alkaline phosphatase less than 2 times ULN
* Lactic dehydrogenase less than 2 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* HIV negative
* No active uncontrolled bacterial, viral, or fungal infection
* No nonmalignant systemic disease that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior irinotecan

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy except small-port radiotherapy for local control
* No concurrent radiotherapy except small-port radiotherapy for local disease control (e.g., pain relief or impending fracture)

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior major surgery

Other:

* No concurrent anticoagulants except warfarin or subcutaneous heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2002-09 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Creaven, MBBS, PhD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Background] Ramnath N, Creaven PJ, Khushalani N, et al.: Pilot studies of antimetabolites preceeded by irinotecan in advanced solid tumors. [Abstract] Eur J Cancer 38 (Suppl 7): S44-5, 2002.
- [Result] Creaven PJ, Slocum HK, Toth K, et al.: Modulation of 5-fluorouracil by irinotecan in advanced solid tumors: a pilot study. [Abstract] Int J Cancer 100 (Suppl 13): A-O78, 94, 2002.